CLINICAL TRIAL: NCT03120169
Title: Effects of a Three Week Treadmill Versus Cycling Endurance Training on Balance, Gait Performance and Exercise Capacity in Patients With Chronic Obstructive Pulmonary Disease - a Pilot Study
Brief Title: Effects of Treadmill Versus Cycling Endurance Training in Patients With COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Schön Klinik Berchtesgadener Land (Other)
Responsible Party: Principal Investigator, Klaus Kenn, Head physican (department of pneumology), Schön Klinik Berchtesgadener Land
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: treadmill vs. cycling in COPD
Record Dates: First submitted 2017-04-13; First posted 2017-04-19 (Actual); Last update posted 2018-02-15 (Actual); Status verified 2018-02

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; exercise; training; cycling; treadmill; walking; pulmonary rehabilitation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treadmill endurance training (Active Comparator)
  Interventions: Other: treadmill endurance training
- cycling endurance training (Active Comparator)
  Interventions: Other: cycling endurance training

INTERVENTIONS:
Other: treadmill endurance training — n = 15 patients with COPD. Walking intensity will be initially set at 80 percent of 6-minute Walking test Speed with progressive increase in Duration and intensity.
  Arms: treadmill endurance training
Other: cycling endurance training — n=15 patients with COPD. Cycling intensity will initially be set at 60 percent of Peak work rate with progressive increase in Duration and intensity
  Arms: cycling endurance training

SUMMARY:
Aim of this study is to investigate the effects of treadmill versus cycling endurance training on Balance, gait performance and exercise capacity in patients with severe chronic obstructive pulmonary disease. Patients will be recruited during a 3-week inpatient pulmonary rehabilitation program and will be randomized into one of two intervention groups. Walking intensity in the treadmill group will be set at 80 percent of the average speed of the 6-minute walking test. The cycling group will exercise at an intensity of 60 percent according to an Initial incremental cycling test.

Patients will perform 5 to 6 training sessions per week. The total exercise duration will be progressively increased from 10 to 30 minutes. Walking or cycling intensity will also be progressively increased if perceived exertion during exercise is rated below 3 on the modified 10-point Borg scale.

ELIGIBILITY:
Inclusion Criteria:

* COPD Stage III or IV according to the global initiative for chronic obstructive lung disease
* impaired exercise capacity (6 Minute walk distance of less than 70% of the reference values from Troosters et al.)

Exclusion Criteria:

* acute, severe exacerbation of COPD
* carbon dioxide of more than 45 mmHg at rest
* any disabilities that prevent patient form walking or cycling
* Patient is not able to walk 20 meters without any aid (for example rollator)

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-03-30 (Actual); Primary Completion 2017-11-27 (Actual); Study Completion 2017-11-27 (Actual)

PRIMARY OUTCOMES:
Change in step symmetry during 20m walking | measurement on day 1 and 21
  Patients walk 20m while wearing the Mc Roberts move test device (triaxial accelerometer) which performs a gait analysis

SECONDARY OUTCOMES:
Change in balance performance during semi-tandem stance | measurement on day 1 and 21
  patients stand still for 10 seconds on a force platform that measures absolute path length of the center of force.
Change in balance performance during Romberg stance | measurement on day 1 and 21
  patients stand still for 10 seconds on a force platform that measures absolute path length of the center of force.
Change in balance performance during single leg stance | measurement on day 1 and 21
  patients stand still for 10 seconds on a force platform that measures absolute path length of the center of force.
Change in muscle power during counter movement jump | measurement on day 1 and 21
  patients jump on a force platform as high as possible. The Outcome is Watt per Kilogram Body weight
Change in 1 Minute sit to stand test | measurement on day 1 and 21
  Patients try to perform as many repetitions as possible of standing up and sitting down from a chair with crossed arms on a force platform during 1 minute
Change in 5 Repetition sit to stand test | measurement on day 1 and 21
  Patients try to perform 5 repetitions of standing up and sitting down from a chair with crossed arms on a force platform as quick as possible
Change in peak muscle strength | measurement on day 1 and 21
  isometric peak torque of the knee extensor muscles are measured in 90° knee angle
Change in 4 meter gait Speed test | measurement on day 1 and 21
  patients have to walk 4 meters at their usual Speed. Outcome is the average Speed during the 4m walk.
Change in 6-minute Walk test | measurement on day 1 and 21
  the best out of two 6- Minute Walk Tests will be used for analysis
Change in Hospital anxiety and Depression scale | measurement on day 1 and 21
  the Hospital anxiety and Depression scale is a questionnaire that evaluates signs of anxiety or depression

CONTACTS AND LOCATIONS:
Locations (1):
- Schoen Klinik Berchtesgadener Land, Schönau am Königssee, Germany